CLINICAL TRIAL: NCT01217177
Title: A Phase I Study of Oral Administration of mTOR Inhibitor Everolimus (RAD001) in Association With Cisplatin and Radiotherapy for the Treatment of Locally Advanced Cervix Cancer
Brief Title: A Study of mTOR Inhibitor Everolimus (RAD001) in Association With Cisplatin and Radiotherapy for Locally Advanced Cervix Cancer
Acronym: PHOENIX I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C24128
Record Dates: First submitted 2010-10-06; First posted 2010-10-08 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Locally Advanced Cervical Cancer
Keywords: Cervical cancer,; radiotherapy,; chemotherapy,; rad001,; everolimus
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Everolimus

ARMS (3):
- 2.5 mg everolimus + radiotherapy + cisplatin (Experimental): patients treated with daily doses of everolimus (2.5mg) in association with radiotherapy and cisplatin (40 mg/m2 of body surface per week, 5 cycles during radiotherapy)
  Interventions: Drug: everolimus
- 5.0 mg everolimus + radiotherapy + cisplatin (Experimental): patients treated with daily doses of everolimus (5.0mg) in association with radiotherapy and cisplatin (40 mg/m2 of body surface per week, 5 cycles during radiotherapy)
  Interventions: Drug: everolimus
- 10 mg everolimus + radiotherapy + cisplatin (Experimental): patients treated with daily doses of everolimus (10mg) in association with radiotherapy and cisplatin (40 mg/m2 of body surface per week, 5 cycles during radiotherapy)
  Interventions: Drug: everolimus

INTERVENTIONS:
Drug: everolimus
  Other Names: RAD001

SUMMARY:
The cervix cancer is the second malignant neoplasia more common between women. The combined treatment involving chemotherapy and radiotherapy was defined as the standard. This study will evaluate the safety, toxicity and maximal tolerated dose (MTD) of everolimus in association with cisplatin and pelvic radiotherapy, in patients with squamous cells carcinoma of uterine cervix, in stages IIB and IIIB.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance of 0, 1 or 2.
2. Evidence of measurable disease of unidimensional form.
3. Epidermoid carcinoma confirmed by histological examination of cervix, stages IIB to IIIB (according to clinical and radiological evaluation), without previous treatment. Absence of positive paraaortic lymph nodes at PET (Positron Emission Tomography).
4. Adequate function of organ, according to following criteria:

   1. Serum levels of aspartate aminotransferase (ASAT/AAT/AST) and alanine aminotransferase (ALT) ≤2.5 x ULN (Upper Limit of Normal)
   2. Total serum bilirubin ≤1.5 ULN
   3. Absolute neutrophils counting ≥1.500/mm3
   4. Platelet counting ≥100.000/mm3
   5. Hemoglobin ≥10.0 g/dL
   6. Serum calcium ≤12.0 mg/dL
   7. Serum creatinine ≤1.5 x ULN and estimate creatinine clearance (Cockroft-Gault) ≥60 mL/min
   8. Prothrombin time ≤1.5 x ULN Obs.: The serum levels of potassium, magnesium, sodium and calcium outside normality range should be corrected before the administration of the first dose of investigational product.
5. Patients with at least one measurable lesion in the baseline period, according to criteria RECIST, version 1.1.
6. Adequate lipid profile: total cholesterol <300 mg/dL and triglycerides <200 mg/dL.
7. Willingness to follow the treatment plan, scheduled visits, laboratory and radiological examinations, as well as other procedures.
8. Signed and dated informed consent form, indicating that the patient (or his/her representative) has received information about all relevant study aspects, before his/her inclusion.

Women with possibility to become pregnant should present a negative serum examination for pregnancy, done within the period of 7 days before the administration of study treatment; and should be willing to use a contraceptive method along the entire study, and for 3 months after the last administration of investigational drug.

Exclusion Criteria:

1. Major surgery <4 weeks before study treatment starting.
2. Any malignant neoplasia in the last 5 years, except for adequately treated melanoma skin cancer.
3. Metastases in the initial diagnostic evaluation [thorax and abdomen computerized tomography (with contrast), pelvis magnetic resonance and PET scanning].
4. Occurrence of some of the following events, during the period of 12 months previously to study medication administration: unstable angina pectoris, symptomatic congestive heart failure (II, III, IV of NYHA), myocardium infarction, severe uncontrolled cardiac arrhythmia, cerebrovascular accident.
5. Positive serology for HIV infection.
6. Patients with positive examinations for hepatitis B (HBsAg, anti-HBs without previous vaccination against HBV and anti-HBc) and hepatitis C (HCV RNA detectable by PCR).
7. Any psychologic, familial, social or geographic problem that could embarrass the adhesion to protocol and study scheme.
8. Patients using other agents under investigation or receiving investigational medications ≤4 weeks before the study treatment starting.
9. Patients presenting some severe and/or uncontrolled medical problem, or other disturbances that could affect their participation in the study, such as, for instance:

   * Unstable angina pectoris, symptomatic congestive heart failure (II, III, IV of NYHA), myocardial infarction ≤12 months before the first administration of study medication, severe uncontrolled cardiac arrhythmia, cerebrovascular accident ≤12 months before the starting of study medication administration;
   * Severely compromised pulmonary function defined by spirometry with 50% of anticipated normal value or decompensated pulmonary disease.
   * Uncontrolled diabetes satisfactorily defined by a fast glycemia result >2.0 x ULN;
   * Any active or uncontrolled disease/infection (acute or chronic) compromising the patient evaluation capability or impeding him/her to complete the study.
   * Hepatic disease with cirrhosis, decompensated hepatic disease, active chronic hepatitis, or persistent chronic hepatitis.
   * Compromising of gastrointestinal (GI) function, or GI disease that could significantly alter the everolimus absorption.
10. Patients unwilling or unable to accomplish the protocol requirements.
11. Hypersensitivity to everolimus or any of its excipients, or to other rapamycins (for instance: sirolimus, temsirolimus).
12. Patients receiving systemic immunosuppressive agents chronically. Inhaling or topic corticosteroids are acceptable. The patients should be receiving stable chronic (not increased within the last month) doses of corticosteroids, with the maximal dose corresponding to 20 mg de prednisone or 10 mg of dexamethasone per day.

Pregnant (that is, having positive examination for beta human chorionic gonadotropin) or lactating women.

Other protocol-defined inclusion/exclusion criteria may apply

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
The toxicity criteria will be evaluated according to National Cancer Institute - Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 3.0. | 12 month

SECONDARY OUTCOMES:
The objective response rate will be evaluated according to clinical/gynecological examination and inconformity with the RECIST criteria (Response Evaluation Criteria in Solid Tumors, version 1.1) | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Brazil (2):
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Rio de Janeiro